CLINICAL TRIAL: NCT01940783
Title: Assessment of the AB HiFocusTM Mid Scala Electrode Movement Using Cone Beam Imaging Following Cochlea Implantation
Acronym: ABMS1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Advanced Bionics (Industry)
Responsible Party: Principal Investigator, Guido Dees, MD, MSc, Maastricht University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL44381.068.13/METC 13-1-054
Record Dates: First submitted 2013-09-09; First posted 2013-09-12 (Estimated); Last update posted 2013-09-12 (Estimated); Status verified 2013-09

CONDITIONS: Cochlear Implantation; Cone-Beam Computed Tomography
MeSH Terms: interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intervention (Other): All participants in the study will receive one pre-operative MRI, prior to cochlear implantation, and two cone-beam computed tomography scans, after cochlear implantation
  Interventions: Radiation: Cone Beam Computed Tomography (CBCT); Device: Magnetic Resonance Imaging (MRI)

INTERVENTIONS:
Radiation: Cone Beam Computed Tomography (CBCT) — Two postoperative CBCT scans, the first one on the day after cochlear implantation and the second after 3 months.
Device: Magnetic Resonance Imaging (MRI) — One pre-operative (before cochlear implantation) MRI scan of the cochlea.

SUMMARY:
One of the contributing factors to the variability in outcomes amongst Cochlear Implant (CI) recipients was reported to be the placement of the electrode array in the scala tympani. It seems that the correct placement of the electrode initially into the scala tympani and subsequent avoidance of dislocation into the scala vestibuli as the insertion progresses, is a key factor in achieving good speech perception outcomes. Another important aspect related to the performance is the achievement of consistent electrical coverage with the electrode. Data reported for electrodes of different manufacturers give depths ranging from 240 - 600 degrees showing the considerable variation across subjects. The HiFocus mid scala electrode was developed to cover one and a quarter turn and with the pre-curved design to be less susceptible to variations in individual cochlea dimensions and insertion techniques. A further mechanical feature of the pre-curved design is the avoidance of forces against the cochlear lateral wall and associated lower susceptibility of the electrode for moving out of the cochlea following insertion. Recently, a cone beam CT (CBCT) technique is being explored in the field of ENT with the potential to overcome some of the issues associated with the conventional CT techniques such as scattering, radiation and low isometric resolution. Images with comparable details to those of e.g. micro CTs are possible with much lower radiation dose. Modern imaging software i.e. 3D Slicer (www.slicer.org) may be used for 3D reconstruction, post processing and Brainsfit for registration. Registration is the alignment of two scans in the same coordinate system. This enables the identification of differences between two images recorded at time x and y. Once accurately superimposed any difference between the two images may be identified with an accuracy of 0.2 mm. Using these methods, one can assess the stability and the position of the electrode in the cochlea.

Objective: The primary objectives of this study are to evaluate the feasibility of using cone beam CT technique in combination with (high resolution) MRI to identify electrode movements following cochlear implant surgery and identify the inter-scalar position of the HFms electrode. The secondary objective is to quantify the average insertion depth and variations of the HFms electrode

ELIGIBILITY:
Inclusion Criteria:

* Adults 18y or older meeting the conventional Dutch CI criteria
* The patient will receives the HiFocus Mid Scala electrode
* No cochlear or neural abnormalities that could compromise the placement of the electrode as assessed by the CI surgeon

Exclusion Criteria:

* Physical or non-physical contraindications for MRI or CT imaging
* No additional disabilities that may prevent active participation and testing as per protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2013-09; Primary Completion 2014-09 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
movement of the electrode post-operatively in millimetres | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert Stokroos, MD PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands